CLINICAL TRIAL: NCT05773690
Title: Effects of a Home-based Quality of Movement Protocol on Functional Movement, Postural Control and Muscular Strength in Obese Subjects
Brief Title: Home-based Training in Obese Individuals
Acronym: FITOB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43C001
Record Dates: First submitted 2023-02-22; First posted 2023-03-17 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obesity
Keywords: Obesity; Functional performance; Postural control; Muscular strength
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Movement Quality group (Experimental): movement quality training based on mobility, stability and motor control exercises
  Interventions: Other: Movement quality
- Conventional resistance training group (Experimental): traditional strength training exercises
  Interventions: Other: Conventional Resistance Training

INTERVENTIONS:
Other: Movement quality — 6-week-home-based training protocols designed to improve general fitness levels and postural control performed in a circuit-training mode (time of work per set 30 s, time of rest between each exercise 15 s, time of rest between sets 2 min, total volume 3 sets) for a duration of 45 min with a frequency of 3 days per week while performing mobility, stability and motor control exercises.
  Arms: Movement Quality group
Other: Conventional Resistance Training — 6-week-home-based training protocols designed to improve general fitness levels and postural control performed in a circuit-training mode (time of work per set 30 s, time of rest between each exercise 15 s, time of rest between sets 2 min, total volume 3 sets) for a duration of 45 min with a frequency of 3 days per week while performing traditional strength training exercises
  Arms: Conventional resistance training group

SUMMARY:
Generally, the enhancement of physical fitness depends on the optimal modulation of different physiological, technical or psychological stimuli and within the factors the would contribute to a decrease performance level, obesity is one of them. In this context, ample evidence shows that obesity is associated with an augmented cardio-metabolic risk, lowered postural control, functional performance and strength-related variables. International guidelines suggests to counteract obesity to respect a minimum dosage of 150 min a week of physical activity at moderate intensity performed with resistance training exercises with a frequency of 2-3 days/week. However, in the aforementioned guidelines there is a little consideration for what concern the quality of motor execution (i.e., "how" an individual performs each movement pattern). In addition, the available literature demonstrates the effectiveness of a "movement-quality" training intervention on fitness parameters and postural control, compared to a mere conventional exercise, in normal-weight individuals . In account to this, the purpose is to evaluate whether a quality of movement protocol would be more effective than a traditional strength training exercise in improving postural control and fitness parameters in subjects with obesity.

ELIGIBILITY:
Inclusion Criteria:

* physical activity frequency at least 1 days per week
* BMI index more than 30 kg/m2
* informed consent signature

Exclusion Criteria:

* aged more than 70 years
* patients with knee pain (Visual Analogue Scale > 7 a.u.)
* history of hip or knee replacement
* severe hip or knee osteoarthrosis
* cardiac or neurological condition contraindicating physical activity

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline functional performance at six weeks | Up to six weeks
  Functional performance using the Functional Movement Screen protocol in arbitrary units with a 0-12 point scale in which higher scores mean a better outcome
Change from baseline body balance at six weeks | Up to six weeks
  Body stability using the modified version of the Balance Error Scoring System protocol in arbitrary units with a 0-30 point scale in which lower scores mean a better outcome
Change from baseline upper-body muscular strength at six weeks | Up to six weeks
  Maximal isometric grip strength in kilograms using the handgrip dynamometer
Change from baseline lower-body muscular strength at six weeks | Up to six weeks
  Amount of time in seconds during a chair raise using the Five Repetition Sit-To-Stand protocol
Change from baseline breathing pattern at six weeks | Up to six weeks
  Breathing pattern performance using the Total Faulty Breathing Scale protocol in arbitrary units with a 0-12 point scale in which lower scores mean a better outcome

SECONDARY OUTCOMES:
Change from baseline weight at six weeks | Up to six weeks
  Body weight using a calibrated weight scale in kilograms
Change from baseline height at six weeks | Up to six weeks
  Body height using a calibrated stadiometer in meters
Change from baseline waist circumference at six weeks | Up to six weeks
  Waist circumference using a 200 centimeters tape measure in centimeters
Change from baseline fat mass at six weeks | Up to six weeks
  Fat mass percentage measurement using a bioelectric impedance analysis

CONTACTS AND LOCATIONS:
Overall Officials: Luca Cavaggioni, Principal Investigator — Istituto Auxologico Italiano IRCCS
Locations (1):
- Istituto Auxologico Italiano IRCCS, Milan, Italy

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26594181/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/15181027/
- See also: Related Info — http://dx.doi.org/10.1016/S0140-6736(05)67483-1
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/26667010/
- See also: Related Info — https://link.springer.com/article/10.1007/s13679-012-0018-7
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30326791/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/11740312/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/25763518/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/30040032/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31500505/